CLINICAL TRIAL: NCT00239590
Title: Effects of Chronic Testosterone on Myocardial Ischaemia and Endothelial Function in Men With Documented Coronary Heart Disease
Brief Title: Testosterone and Myocardial Perfusion in Coronary Heart Disease (CHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Organon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000AE13B
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy dispensing of study medication that was randomized by supplier
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone (Experimental): oral testosterone undecanoate, 80mg twice daily (Andriol Testocaps, Organon, The Netherlands) for 8 weeks
  Interventions: Drug: Testosterone undecanoate
- Placebo (Placebo Comparator): identical to active medication, taken in an identical way to the active arm
  Interventions: Drug: Testosterone undecanoate

INTERVENTIONS:
Drug: Testosterone undecanoate — Licensed for androgen deficiency
  Other Names: Andriol; Org 538

SUMMARY:
Testosterone has traditionally been regarded as a risk factor for heart disease due to the fact that males have a higher incidence of this disease than women, at least until the menopause. However recent studies have shown that men with low levels of testosterone may be at an increased risk of developing coronary heart disease (furring up of the blood vessels supplying blood to the heart). Our group has demonstrated a relaxing effect of testosterone in isolated animal coronary arteries (blood vessels supplying blood to the heart). We have shown that short-term testosterone administration can increase coronary artery and brachial artery (blood vessel in the arm) blood flow and can decrease the lack of blood supply to the heart muscle in men with coronary artery disease. These findings indicate a need for similar but longer-term studies to investigate the possible beneficial effects of longer-term testosterone therapy on the heart and blood vessels. Should this treatment be shown to be beneficial to men with coronary artery disease it may be a useful additional therapy for men with the furring up of arteries in the heart and the resulting angina.

Aim To investigate our hypothesis that testosterone can beneficially affect myocardial perfusion, vascular reactivity, metabolic risk factors for coronary heart disease and improve quality of life in men with low plasma testosterone levels and coronary heart disease.

DETAILED DESCRIPTION:
The main purpose of this project is to determine whether testosterone treatment over a number of weeks can beneficially affect myocardial perfusion, vascular reactivity, metabolic risk factors and quality of life in men with documented coronary heart disease. Men with documented significant coronary artery disease and a positive exercise test for myocardial ischaemia will be enrolled into the study. They will be randomised to active testosterone therapy (5 mg/day) or placebo for 2 months. After 2 months they will undergo MRI perfusion scanning, radial artery applanation tonometry to assess endothelial function, blood sampling for analysis of metabolic risk factors for coronary heart disease, complete quality of life questionnaires and will cross-over to the opposite treatment. After a further 2 month period these tests will be repeated. Angina diaries will be kept for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged 35 to 75 years
* Angiographically proven coronary artery disease (70 percent lesion in at least one major coronary artery, or major branch), including patients post-coronary artery bypass graft (CABG) and percutaneous coronary intervention (PCI)
* Plasma testosterone less than or equal to 12 nmol/l
* Normal prostate specific antigen (PSA; normal range 0 - 4 g/l)
* Willing to give written informed consent

Exclusion Criteria:

* Significant arrhythmia, particularly those which would affect interpretation of the ST-segment of the ECG
* Treatment with digitalis
* Treatment with testosterone or similar hormonal therapy
* Thoracic or abdominal surgery within the previous 3 months
* Haemoglobin >16 g/dL
* Haematocrit >50 percent
* History of hormone-dependent cancer such as prostate or breast cancer
* Hypercalcaemia
* Nephrosis
* Pacemaker or automated implantable cardiac defibrillator
* Implanted ferromagnetic arterial clips
* Left ventricular hypertrophy
* New York Heart Association (NYHA) III or IV functional class
* Intolerance of confined spaces
* Previous allergic reaction to Gadolinium
* Participation in another research study within the previous 60 days
* Unwilling to give written informed consent

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2004-04-24 (Actual); Study Completion 2004-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Collins, MA MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Trust, London, United Kingdom

REFERENCES:
- [Result] Webb CM, Elkington AG, Kraidly MM, Keenan N, Pennell DJ, Collins P. Effects of oral testosterone treatment on myocardial perfusion and vascular function in men with low plasma testosterone and coronary heart disease. Am J Cardiol. 2008 Mar 1;101(5):618-24. doi: 10.1016/j.amjcard.2007.09.114. Epub 2007 Dec 21. PMID 18308009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients at a tertiary referral NHS hospital in London, UK. Eligible patients were invited to participate by post. Interested participants returned an eligibility questionnaire. Those fulfilling the inclusion/exclusion criteria were invited to attend for a screening/consent appointment.
Pre-assignment Details: Blood was taken at a screening visit. Those not fulfulling the inclusion/exclusion criterial were excluded.
Groups:
- Testosterone (First, Then Placebo): oral testosterone undecanoate, 80mg twice daily (Andriol Testocaps, Organon, The Netherlands) for 8 weeks.
  At the end of 8 weeks, patients were evaluated, then crossed-over to placebo for 8 weeks. No wash-out period.
  Testosterone undecanoate: Licensed for androgen deficiency
- Placebo (First, Then Testosterone): identical to active medication, taken in an identical way to the active arm for 8 weeks.
  At the end of the 8 week placebo treatment phase evaluation visit, patients crossed-over to the testosterone treatment arm for 8 weeks. No wash-out period.
Period: Randomized
Arm/Group | Testosterone (First, Then Placebo) | Placebo (First, Then Testosterone)
Started | 14 | 14
Completed | 14 | 12
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Started Intervention After Randomization
Arm/Group | Testosterone (First, Then Placebo) | Placebo (First, Then Testosterone)
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0
Period: Completed Study Protocol
Arm/Group | Testosterone (First, Then Placebo) | Placebo (First, Then Testosterone)
Started | 14 | 12
Completed | 13 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 28 participants were randomized to testosterone or placebo first then crossed over after 8 weeks, and 25 patients completed the study protocol. There was no carry-over effect detected from the first to the second period, therefore the data presented here are pooled data of both treatment arms.
Groups:
- All Study Participants: All participants randomized to study medication (n=28), whether randomized to testosterone or placebo first.
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion
Description: Myocardial perfusion (blood flow in the heart muscle) in subendocardial myocardial segments (one of the inner layers of heart muscle), supplied by coronary arteries without significant obstruction. This was measured using Cardiovascular Magnetic Resonance (CMR) imaging and a dual-bolus gadnolinium infusion protocol.
  Myocardial perfusion index = the ratio between myocardial perfusion measurements following adenosine-induced stress and rest measurements.
Time Frame: Testosterone versus placebo (8 week treatment period)
Population: 22 patients had assessable CMR data for both evaluation visits.
Measure: Mean (Standard Deviation); unit: myocardial perfusion index
Groups:
- Testosterone: Pooled first and second treatment phase data.
  oral testosterone undecanoate, 80mg twice daily (Andriol Testocaps, Organon, The Netherlands) for 8 weeks.
  Testosterone undecanoate: Licensed for androgen deficiency
- Placebo: pooled first and second treatment phase data
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 22 | 22
myocardial perfusion index | 1.83 (0.9) | 1.52 (0.65)

2. Secondary Outcome: Endothelial Function
Description: The endothelium is a single layer of cells that line all blood vessels and regulates arterial function. Coronary artery disease causes dysfunction of the endothelium but some substances/drugs help to reverse this dysfunction. In this study, endothelial function was measured by radial applanation tonometry which measures the blood pressure waveform during each cardiac cycle (heart beat). Radial artery pulse recordings were acquired, with an averaged waveform generated from 20 sequential waveforms. Augmentation index (AIx) is derived from this averaged waveform, and is the ratio of the pulse pressure at the second systolic arterial pressure waveform peak to that of the first systolic peak. The change in AIx before and after salbutamol (400mcg) is a measure of endothelial function.
Time Frame: Testosterone versus placebo (8 week treatment period)
Population: A total of 17 patients had endothelial function assessments - the same patients took both interventions in a randomized cross-over design.
Measure: Mean (Standard Deviation); unit: Augmentation index
Groups:
- Testosterone: oral testosterone undecanoate, 80mg twice daily (Andriol Testocaps, Organon, The Netherlands) for 8 weeks
  Testosterone undecanoate: Licensed for androgen deficiency
  Active and placebo given in a cross-over design
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 17 | 17
Augmentation index | 76.5 (9.5) | 79.4 (7.8)

ADVERSE EVENTS:
Time Frame: Event data were collected from time of participant inclusion in the study until the end of the final study visit (end of the second treatment phase and assessment visit) - a total of approximately 20 weeks. There was no formal long-term follow-up.
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=28) | Placebo (N=28)
Hospitalization (Nervous system disorders) | 1 (1) | 0 (0) — Suspected stroke and pneumonia approximately 2 weeks after starting study medication (active arm). Serious adverse event (SAE) not considered to be related to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=28) | Placebo (N=28)
Low mood (Nervous system disorders) | 0 (0) | 1 (1) — Patient complained of general malaise and feeling of exhaustion, 'almost a depression' and stopped the study medication (placebo). He decided to withdraw from the study. These symptoms resolved after 2 weeks off the study medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes